CLINICAL TRIAL: NCT00125918
Title: PHIRST-1: Randomized, Double-Blind, Placebo-Controlled Phase 3 Study of the Phosphodiesterase Type 5 (PDE5) Inhibitor Tadalafil in the Treatment in Patients With Pulmonary Arterial Hypertension
Brief Title: PHIRST-1: Tadalafil in the Treatment of Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ICOS Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10303; H6D-MC-LVGY
Record Dates: First submitted 2005-08-01; First posted 2005-08-02 (Estimated); Last update posted 2008-02-21 (Estimated); Status verified 2008-02

CONDITIONS: Pulmonary Hypertension
Keywords: Hypertension, Pulmonary; Pulmonary Heart Disease
MeSH Terms: conditions — Hypertension, Pulmonary; Hypertension; Pulmonary Heart Disease | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: placebo
- 2 (Active Comparator): 2.5 mg tadalafil
  Interventions: Drug: tadalafil
- 3 (Active Comparator): 10 mg tadalafil
  Interventions: Drug: tadalafil
- 4 (Active Comparator): 20 mg tadalafil
  Interventions: Drug: tadalafil
- 5 (Active Comparator): 40 mg tadalafil
  Interventions: Drug: tadalafil

INTERVENTIONS:
Drug: tadalafil — tadalafil 2.5 mg and placebo tablets taken by mouth once a day for 16 weeks.
  Other Names: LY450190; Cialis; IC351
  Arms: 2
Drug: tadalafil — tadalafil 10 mg and placebo tablets taken by mouth once a day for 16 weeks.
  Other Names: LY450190; Cialis; IC351
  Arms: 3
Drug: tadalafil — tadalafil 20 mg and placebo tablets taken by mouth once a day for 16 weeks.
  Other Names: LY450190; Cialis; IC351
  Arms: 4
Drug: tadalafil — tadalafil 40 mg and placebo tablets taken by mouth once a day for 16 weeks.
  Other Names: LY450190; Cialis; IC351
  Arms: 5
Drug: placebo — placebo tablet taken by mouth once a day for 16 weeks
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of tadalafil for the treatment of pulmonary arterial hypertension.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter study. The key measure of effectiveness of the study drug will be determined using a 6-minute walk test. Eligible patients will be treated for 16 weeks and may be eligible to enter a 52-week extension phase study (PHIRST-2). Study procedures for both studies (PHIRST-1 and PHIRST-2) will include routine blood tests, medical history, physical exams, questionnaire responses, and exercise tests.

ELIGIBILITY:
Inclusion Criteria:

* At least 12 years of age.
* Body weight at least 40 kg (approximately 88 pounds).
* Pulmonary hypertension (PAH) that is either idiopathic; related to collagen vascular disease; related to anorexigen use; associated with an atrial septal defect (resting SaO2 greater than or equal to 88%); with surgical repair, of at least 1 year duration, of a congenital systemic-to-pulmonary shunt.
* If on bosentan, must be at the maximal dose of 125 mg twice daily for a minimum of 12 weeks prior to screening and have an AST/ALT less than 3 times normal.
* History of PAH established by a resting mean pulmonary artery pressure greater than or equal to 25 mm Hg, pulmonary artery wedge pressure less than or equal to 15 mm Hg, and pulmonary vascular resistance greater than or equal to 3 Wood units via right heart catheterization
* Have World Health Organization functional class I, II, III or IV status.
* Have a qualifying 6-minute walk test distance at screening
* Have no evidence of significant parenchymal lung disease

Exclusion Criteria:

* Are nursing or pregnant.
* PAH due to conditions other than noted in the above inclusion criteria.
* History of left-sided heart disease.
* History of atrial septostomy within 3 months before study entry
* History of angina pectoris or other condition that was treated with long-or short-acting nitrates within 12 weeks before administration of study drug.
* History of symptomatic coronary disease.
* Have any therapy with a prostacyclin or analogue, L-arginine, phosphodiesterase (PDE) inhibitor, or investigational drug within 4 weeks before administration of study drug.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2005-08; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
6 minute walk distance change from baseline to Week 16 | 16 weeks

SECONDARY OUTCOMES:
World Health Organization (WHO) functional class, Borg dyspnea, cardiopulmonary hemodynamics, quality of life - change from baseline to Week 16 | 16 weeks
Time to first occurrence of clinical worsening | Not defined

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
- France (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vandœuvre-lès-Nancy
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bergamo, Italy

REFERENCES:
- [Derived] Ferguson-Sells L, Velez de Mendizabal N, Li B, Small D. Population Pharmacokinetics of Tadalafil in Pediatric Patients with Pulmonary Arterial Hypertension: A Combined Adult/Pediatric Model. Clin Pharmacokinet. 2022 Feb;61(2):249-262. doi: 10.1007/s40262-021-01052-8. Epub 2021 Aug 11. PMID 34379314
- [Derived] Galie N, Brundage BH, Ghofrani HA, Oudiz RJ, Simonneau G, Safdar Z, Shapiro S, White RJ, Chan M, Beardsworth A, Frumkin L, Barst RJ; Pulmonary Arterial Hypertension and Response to Tadalafil (PHIRST) Study Group. Tadalafil therapy for pulmonary arterial hypertension. Circulation. 2009 Jun 9;119(22):2894-903. doi: 10.1161/CIRCULATIONAHA.108.839274. Epub 2009 May 26. PMID 19470885
- See also: The Pulmonary Hypertension Association (PHA) is an organization that provides support, education, advocacy, and awareness about pulmonary hypertension. — http://www.phassociation.org
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com